CLINICAL TRIAL: NCT07218419
Title: Comparison of Methods for Assessing Intraocular Lens Position
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MDEV109TDMD
Record Dates: First submitted 2025-10-07; First posted 2025-10-20 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Tilt and Decentration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- IOL Decentration: The objective is to evaluate two methods for assessing IOL tilt and decentration in patients who have been unilaterally or bilaterally implanted with a refractive or diffractive non- toric TECNIS IOL before participating into this study. The agreement will be assessed between the decentration measurements derived from retro-illuminated slit lamp image analysis and those obtained from the subjective slit lamp grading method.
  Interventions: Diagnostic Test: IOL Decentration Assessment

INTERVENTIONS:
Diagnostic Test: IOL Decentration Assessment — This study assesses two methods to measure IOL decentration. Each subject will be evaluated in only one eye with both methods for assessing IOL decentration:
  (i) retro-illuminated slit lamp image analysis (objective slit lamp method) and (ii) subjective slit lamp grading method. There is no treatment or intervention on this study.
  Other Names: Basic Science

SUMMARY:
Prospective, multi-center, non-interventional, open label, clinical study.

DETAILED DESCRIPTION:
The objective is to evaluate two methods for assessing IOL tilt and decentration in patients who have been unilaterally or bilaterally implanted with a refractive or diffractive nontoric TECNIS IOL before participating into this study. The agreement will be assessed between the decentration measurements derived from retro-illuminated slit lamp image analysis and those obtained from the subjective slit lamp grading method.

ELIGIBILITY:
Inclusion:

All criteria apply to study eye.

The subject must:

* Read, understand, and sign the informed consent and HIPAA authorization forms, and receive a fully executed copy of the signed forms.
* Appear capable and willing to adhere to the clinical protocol procedures.
* Be 22 years of age or older at the time of screening.
* Have undergone unilateral or bilateral implantation with a desired TECNIS non-toric IOL design (e.g., refractive or diffractive).
* Be at least three months postoperative in the study eye.

Exclusion:

All criteria apply to study eye.

The subject must NOT:

* Any medical or ocular history, in the opinion of the investigator, that may impact study procedures such as ocular trauma, pseudoexfoliation syndrome, retinal pigment degeneration, macular pathology, glaucoma, retinal disease, corneal disease, or corneal opacities.
* Have any condition that may affect the eye's ability to fixate (e.g., amblyopia).
* Have a history of corneal or intraocular surgery other than cataract surgery.
* Be using ocular or systemic medications known to interact with dilation drops.
* Have a history of hypersensitivity, allergic reaction or other contraindication to dilation drops.
* Have clinically significant pupil abnormalities (e.g., non-reactive, fixed, or abnormally shaped pupils).
* Have an intraocular pressure of ≥ 21mm Hg before mydriasis.
* Have a mydriatic pupil diameter of less than 6mm.
* Have participated in clinical trial within 7 days prior to study enrollment.
* Be an employee (e.g., Investigator, Coordinator, or Technician) or immediate family member (including partner, child, parent, grandparent, grandchild, or sibling) of an employee of the clinical site or study sponsor.
* Be currently pregnant or lactating.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants eligible for the study must be 22 years of age or older and have received a refractive or diffractive nontoric TECNIS IOL in at least one eye. Additionally, they must be at least three months post-operative in the designated study eye. The Investigator should choose the eye without any clinically significant medical conditions that may interfere with the evaluation of IOL tilt and decentration using the testing methods specified in this study. If both eyes meet the eligibility criteria, the right eye will be designated as the study eye.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-01-16 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
IOL Decentration | 3 months
  * Magnitude of Decentration relative to the center of the pupil.
  * Direction of Decentration relative to the center of the pupil

CONTACTS AND LOCATIONS:
Overall Officials: Surgical Vision Inc. Johnson and Johnson, Study Director — Study Director
Locations (2):
- United States (2):
  - Empire Eye & Laser Center, Bakersfield, California
  - Jones Eye Center, Sioux City, Iowa

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu